CLINICAL TRIAL: NCT05944185
Title: Phase I/II Study of αPD1-MSLN-CAR T Cells in MSLN-positive Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Cell Therapy Group Co.,Ltd (Industry)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BZDS1901-CTP-I/II-01
Record Dates: First submitted 2023-07-06; First posted 2023-07-13 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR T cells (Experimental)
  Interventions: Drug: αPD1-MSLN-CAR T Cells

INTERVENTIONS:
Drug: αPD1-MSLN-CAR T Cells — αPD1-MSLN-CAR T Cells

SUMMARY:
An open, multicenter, phase I/II study to evaluate the safety, tolerability, and effectiveness of αPD1-MSLN-CAR T cells in patients With MSLN-positive advanced solid tumors

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histological or cytological diagnosis of advanced solid tumors#
* Patients must have failed established standard medical anti-cancer therapies#
* Greater than or equal to 18 years of age and less than or equal to 70 years of age on day of signing informed consent#
* Life expectancy >3 months#
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or
* Subjects must meet blood coagulation parameters and have adequate venous peripheral access for apheresis. Patients must also have adequate mononuclear cells for CAR T cell manufacturing#
* Staining of MSLN must be greater than 50% of the cells in the tumor tissue and with apparent expression in the membrane. PD-L1 expression must be positive. Tissue obtained for the biopsy must be ≤1 year prior to enrollment for screening, not have been previously irradiated or exposed to chemotherapy. If unavailable, new tissue material from a recently obtained surgical or diagnostic biopsy is mandatory for this trial#
* Satisfactory organ and bone marrow function as defined by the following:

  1. Adequate bone marrow function in the opinion of the Investigator for lymphocyte-depleting chemotherapy: absolute neutrophil count must be greater than ≥ 1.5×109/L, lymphocyte count must be greater than ≥ 0.5×109/L, platelets must be greater than ≥ 90×109/ L, hemoglobin must be greater than ≥ 90g/L without transfusion within 7 days or dependency on EPO;
  2. Total bilirubin must be less than or equal to two times (≤2.0x) the institutional normal upper limit; transaminases, serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST), must be less than or equal to 2.5 times (≤2.5x) the institutional normal upper limit (≤2.5x if there is hepatic metastasis);
  3. Creatinine must be less than or equal to one and one half times (≤ 1.5x) the institutional normal upper limit or eGFR ≥ 60ml/ min/1.73m^2 [eGFR=186×#age#-0.203×SCr-1.154#mg/dl#,for female the eGFR shoud be timed by 0.742];
  4. International normalized ratio (INR) or the PT is not greater than one and one half times (≤ 1.5) the upper limit of normal;
  5. Lung function: ≤ CTCAE grade 1 dyspnea and SaO2≥ 91%
  6. Cardiac function: cardiac ejection fraction (LVEF) must be greater than fifty percent (≥50%) by echocardiogram or MUGA one month before enrollment.
* Subjects must have measureable disease as defined by RECIST 1.1 criteria;
* Subjects sufficiently understand the trial and willingly sign the informed consent;

  - Page 3 of 5 -
* For concurrent medication:

  1. Systemic therapeutic corticosteroids must be stopped 72 hours before CAR-T infusion. However, patients using physiologic replacement doses of corticosteroids, or its equivalent, will be considered eligible;
  2. Immunosuppressive therapy must be stopped within four (4) weeks prior to enrollment;
* Male and Female subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for at least 12 months following the last dose of the study cell infusion and until no CAR-T cells can be detected after two consecutive PCR tests.

Exclusion Criteria:

* Prior therapy with targeted therapy or cell therapy against MSLN#
* Prior therapy with any gene therapy (including CAR-T cell therapy) or any T cell therapy home and abroad#
* Active bacteria, viral or fungal infection, and not contained after antiinfective therapy (positive results in the blood ≤72 hours before infusion);
* Patient is positive for Syphilis, Human Immunodeficiency Virus (HIV) , active Hepatitis B (HBsAg reactive) or Hepatitis C (HCV RNA (qualitative) is detected);
* Patient has a medical condition such as autoimmune disease or organ transplantation that requires chronic systemic steroid therapy or requires any other form of immunosuppressive medication;
* History of severe cardiac or pulmonary disease, including hypertension that cannot be controlled by medication, and any of the conditions occurred within the past 6 months: congestive heart failure (New York Heart Association functional classification ≥3), cardiac angioplasty and stents, myocardial infarction, unstable angina, or other clinically significant heart disease#
* Detectable clinically relevant central nervous system (CNS) metastases and/or pathology such as epilepsy/seizure, brain Ischemia/ hemorrhage, dementia, cerebellar disease, or autoimmune disease affecting central nervous system#
* Patient has a history or current evidence of any condition such as neurotic, psychiatric, immune, metabolic and infectious disease, on any therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study, or is not in the best interest of the patient to participate, in the opinion of the treating Investigator#
* Patient has a known history of a hematologic malignancy, or of another malignant primary solid tumor concurrently, with the exception of :

  1. Patients with in situ cervical cancer or breast cancer with no evidence of disease for ≥ 3 years after curative treatments;
  2. Patients who underwent successful definitive resection of in situ cancer with no evidence of disease for ≥5 years;
* Has had chemotherapy, radioactive, small molecules, biological cancer therapy, immunotherapy or other investigational drugs within 4 weeks prior to the initiation of the study#
* Pregnant or breastfeeding women;
* Investigators think that patient has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the patient's participation for the full duration of the study and cooperation with the requirements of the trial, uncontrolled medical, psychological, familial, sociological, or geographical conditions, or is not in the best interest of the patient to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Incidence of Treatment Related adverse events (AEs) | Up to 12 months
  Incidence of treatment related AEs, AEs of special interest and serious adverse events(SAEs).
Phase Ib: Identification of Maximum Tolerated Dose (MTD) | day1-day28
  Incidence of dose-limiting toxicities (DLTs)
Phase II: Objective Response Rate (ORR), as assessed by IRC | Up to 12 months
  The Objective Response Rate (ORR) is the percentage of participants who achieved a best overall response of Complete Response (CR) or Partial Response (PR) based on RECIST version 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Jianchun Duan, Principal Investigator — National Cancer Center Cancer Hospital Chinese Academy of Medical Sciences
Locations (1):
- National Cancer Center Cancer Hospital Chinese Academy of Medical Sciences, Beijing, China